CLINICAL TRIAL: NCT05395312
Title: Evaluation of Blended Stepped-care Mental Well-being Intervention for Adults: A Randomized Controlled Trial
Brief Title: Evaluation of Online Mental Well-being Intervention for Working Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Winnie W.S. MAK, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB/REC: 2021.334
Record Dates: First submitted 2022-05-18; First posted 2022-05-27 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Mental Well-being; Mental Health Issue; Mental Health Wellness 1
Keywords: online; stepped-care; mental well-being; working adults; RCT; psychological distress; depression; anxiety
MeSH Terms: conditions — Psychological Well-Being; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Researchers do not know the group allocation until the end of study. An individual party is responsible to randomly allocate participants into blended stepped-care group and waitlist control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blended stepped-care group (Experimental): Participants in the blended stepped-care group can access the online materials at levels based on their psychological distress through login to the platform of the JCTH+ project. They can choose their preferred online courses by using online course taster. Also, they can join offline programs corresponding to their levels of psychological distress.
  Interventions: Other: Online blended stepped-care mental well-being platform
- Waitlist control group (No Intervention): Participants in the waitlist control group will receive their usual treatment and follow their usual practice if any. They will be offered the opportunity to receive the services in the blended stepped-care group after the study has ended.

INTERVENTIONS:
Other: Online blended stepped-care mental well-being platform — Participants in experimental group will be stratified according to their level of anxiety and/or depressive symptoms.
  Level 2 (normal range)
  * Topic-based personal growth articles, exercises, and chatbots
  * Webinars and talks on varied mental health related topics
  * Virtual support community
  Level 3 (mild to moderate)
  * Online self-guided mental well-being training programs, such as mindfulness-based intervention, rumination-focused cognitive behavioural therapy, and transdiagnostic cognitive behavioural therapy
  * Offline/online skills-based workshops, questions-and-answers sessions, retreats
  Level 4 (severe)
  * Online coach-guided mental well-being training programs, such as mindfulness-based intervention, rumination-focused cognitive behavioural therapy, and transdiagnostic cognitive behavioural therapy
  * Offline/online group therapy, 4-week group cognitive behavioural therapy or 8-week group mindfulness-based cognitive therapy
  Arms: Blended stepped-care group

SUMMARY:
This study aims to evaluate the effectiveness and cost-effectiveness of the online stepped-care mental well-being system together with offline programs in comparison to care as usual. This study will provide important findings for future health economic analyses of blended stepped-care mental well-being interventions which may increase public's access to mental well-being services and ease the long waiting time under the current public healthcare system. It is hypothesized that participants in the intervention group show (H1) greater reduction in depressive and anxiety symptoms, (H2) better improvement of well-being, (H3) better improvement of quality of life, and (H4) lower incremental cost-effectiveness ratio (ICER), compared to care as usual.

DETAILED DESCRIPTION:
In Hong Kong, mental disorders such as anxiety and depression are common. With the 13.3% of respondents reported to have symptoms of anxiety, depression, or comorbid anxiety and depression, only 26% of them sought for mental health services within the past year. The same morbidity survey also revealed as much as 11.25% of working adults were affected by symptoms of common mood disorders. The COVID-19 pandemic and social movement further increase stress and feelings of uncertainties on the general population. Two telephone surveys of over 1000 working adults each conducted in Dec 2017 and Feb 2020 suggested that 24.3% and 26.3% of working adults experienced anxiety and depressive symptoms in the past two weeks (the Jockey Club TourHeart Project, JCTH). Yet, 46% and 28% of respondents indicated they would not seek help for their psychological distress.

The services provided by the current public health system and private sector in Hong Kong are insufficient, mainly due to a shortage of professionals such as clinical psychologists and psychiatrists. There are also relatively less resources from the government and non-governmental organizations to the working adults comparing with the more 'vulnerable' populations, such as children, adolescents, and older people. A survey conducted in 2019 found more than 90% of the interviewees expressed that their companies did not offer sufficient support on employees' mental well-being. The same study suggested that 55% of the interviewees reported feeling ashamed about their own mental health issues or knowing someone with mental health issues, with these being named barriers to service. The needs of the working adults are unlikely to be fulfilled by companies or employers because of tightened budget, lack of awareness and knowledge, and stigma on mental illness. There exists a significant gap between the tremendous need for taking care of mental well-being and the mental well-being support services among the working adults in Hong Kong.

Online Stepped-Care Mental Well-being Interventions

The mental well-being services provided by the current public healthcare system in Hong Kong mainly rely on the traditional face-to-face and one-to-one therapy sessions. Due to the shortage of professionals, the waiting time for new service users is unbearably long while the follow-ups for returning users is infrequent. Also, priority is usually given to people with more severe mental well-being issues which causes the waiting time for people with mild to moderate mental well-being needs even longer.

The stepped-care model takes the approach of using the least restrictive method to commensurate with mental well-being needs and profiles of the service users with self-correcting process. Based on timely assessment of mental well-being status of the service users, corresponding treatments with matched levels of intensity could be utilized. According to treatment progress of the service users, stepped-care model enables mechanism to step up or down by adjusting the levels of intensity of the interventions. The National Institute of Health and Care Excellence (NICE) has issued evidence-based guidance detailing the stepped-care model for treatment of depression and anxiety in order to enhance treatment of these common mental disorders. A systematic review and meta-analysis suggested that the stepped-care approach was significantly better than care-as-usual in the treatment of anxiety although it could not significantly prevent or reduce future incidence of depression and anxiety. The stepped-care approach is proposed to reduce time, cost, and associated treatment burden on the clinicians and the service users.

Internet-based interventions for anxiety and depression have been found to be effective in reducing anxiety and depressive symptoms. Transdiagnostic treatments are recommended rather than disorder-specific treatments with the consideration of co-occurrence of depression and anxiety. Internet-delivered cognitive behavioural therapy has been recommended by the NICE guidelines as one of the low-intensity interventions for people with depression and anxiety. Applying the stepped-care model with an online mental well-being self-care platform, the service users can access mental well-being services at any time and any place. Online scientific evidence-based psychological interventions provide solutions for the service users on their mental well-being issues without practical burdens resulted from long waiting time, high expenses, and stigmatization.

Cost-Effectiveness

Cost is one of the elements causing economic burdens of mental disorders. Among the working population, absenteeism and productivity losses added extra costs to the companies. These mental well-being issues costs employers HKD 5.5-12.4 billion a year on average. Data about cost-effectiveness of online stepped-care mental well-being approach was relatively scarce. A systematic review suggested that internet-based therapy has more than 50% probability of being cost-effective compared with no treatment or conventional face-to-face therapy. Results from two studies with randomised controlled trial design found that online therapy was more cost-effective than treatment-as-usual. Some studies suggest that the cost-effectiveness of using stepped-care approach remains inconclusive. There is a need to understand the cost-effectiveness of the online stepped-care mental well-being approach. Economic evaluation is a common way to examine the cost-effectiveness of interventions by estimating the treatment effects relative to the associated cost.

The Current Study

The current study aims to evaluate the effectiveness and cost-effectiveness of the online stepped-care mental well-being system together with offline programs in comparison to the care-as-usual group. This study will provide important findings for future health economic analyses of blended stepped-care mental well-being interventions which may increase public's access to mental well-being services and ease the long waiting time under the current public healthcare system. It is hypothesized that participants in blended stepped-care group will show (H1) greater reduction in depressive and anxiety symptoms, (H2) better improvement of well-being, (H3) better improvement of quality of life, and (H4) lower incremental cost-effectiveness ratio (ICER), compared to the care-as-usual group.

Participants will be recruited through (1) mass mailing and emails to staff through higher educational institutes, unions, enterprises, professional, and nongovernmental organizations, (2) distribution of posters and leaflets to enterprises, governmental organisations, local nongovernmental organisations, social service centres, public libraries, health clinics, counselling centres, (3) information posting at popular online networking platforms (e.g., Facebook and Instagram), newspapers, magazines, roadshows, and promotional booths for recruitment purposes.

Upon obtaining consent of the study, participants will complete a screening. Participants with high suicidal risk will be recommended with appropriate referral services in public and private settings as follow-up after seeking approval from clinical psychologist in the team. Eligible participants will be assigned to blended stepped-care group or care-as-usual group by randomization after completion of baseline questionnaire. Participants in the blended stepped-care group can access the online materials at levels based on their psychological distress through login to the platform of the JCTH+ project. They can choose their preferred online courses by using online course taster. Also, they can join offline programs corresponding to their levels of psychological distress. Participants in the waitlist control group will receive their usual treatment and follow their usual practice if any. They will be offered the opportunity to receive the services in the blended stepped-care group after the study has ended. Both groups of participants will be invited to complete the set of questionnaires online at baseline, 3rd and 6th month.

ELIGIBILITY:
Inclusion Criteria:

* Working adults aged 18 years old or above
* Able to read and understand Chinese, spoken Cantonese
* Have access to the Internet

Exclusion Criteria:

* High suicidal risk
* Who are unwilling to receive the intervention by random assignment
* Existing users of the JCTH project platform
* Non-working adults

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2022-07-30 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms - Patient Health Questionnaire (PHQ-9) | at baseline
  It includes 9 items to assess the extent of which respondents are bothered by depression related symptoms using a 4-point Likert scale from 0 (not at all) to 3 (nearly every day). PHQ-9 has been validated and used widely in the general population for screening and measuring depression severity. Total scores range from 0 to 27. Scores of 5, 10, 15, and 20 denote mild, moderate, moderately severe, and severe level of depression respectively.
Depressive symptoms - Patient Health Questionnaire (PHQ-9) | 3rd month
  It includes 9 items to assess the extent of which respondents are bothered by depression related symptoms using a 4-point Likert scale from 0 (not at all) to 3 (nearly every day). PHQ-9 has been validated and used widely in the general population for screening and measuring depression severity. Total scores range from 0 to 27. Scores of 5, 10, 15, and 20 denote mild, moderate, moderately severe, and severe level of depression respectively.
Depressive symptoms - Patient Health Questionnaire (PHQ-9) | 6th month
  It includes 9 items to assess the extent of which respondents are bothered by depression related symptoms using a 4-point Likert scale from 0 (not at all) to 3 (nearly every day). PHQ-9 has been validated and used widely in the general population for screening and measuring depression severity. Total scores range from 0 to 27. Scores of 5, 10, 15, and 20 denote mild, moderate, moderately severe, and severe level of depression respectively.
Anxiety symptoms - Generalized Anxiety Disorder Assessment (GAD-7) | at baseline
  It is a 7-item scale to assess the extent of which respondents are bothered by anxiety related symptoms using a 4-point Likert scale from 0 (not at all) to 3 (nearly every day). GAD-7 is a well-established scale with good reliability and procedural validity. Total scores range from 0 to 21. Scores of 5, 10, and 15 denote mild, moderate, and severe level of anxiety respectively.
Anxiety symptoms - Generalized Anxiety Disorder Assessment (GAD-7) | 3rd month
  It is a 7-item scale to assess the extent of which respondents are bothered by anxiety related symptoms using a 4-point Likert scale from 0 (not at all) to 3 (nearly every day). GAD-7 is a well-established scale with good reliability and procedural validity. Total scores range from 0 to 21. Scores of 5, 10, and 15 denote mild, moderate, and severe level of anxiety respectively.
Anxiety symptoms - Generalized Anxiety Disorder Assessment (GAD-7) | 6th month
  It is a 7-item scale to assess the extent of which respondents are bothered by anxiety related symptoms using a 4-point Likert scale from 0 (not at all) to 3 (nearly every day). GAD-7 is a well-established scale with good reliability and procedural validity. Total scores range from 0 to 21. Scores of 5, 10, and 15 denote mild, moderate, and severe level of anxiety respectively.

SECONDARY OUTCOMES:
Productivity - The Institute for Medical Technology Assessment (iMTA) Productivity Costs Questionnaire (iPCQ) | at baseline, 3rd, and 6th month
  It is a 12-item scale to assess productivity losses of paid work due to absenteeism and presenteeism, as well as productivity losses related to unpaid work. Calculation of the scale score will be based on iMTA formula.
Medical consumption - Utilization of Health Services | at baseline, 3rd, and 6th month
  It is a questionnaire to assess the medical consumption in the local context of Hong Kong by counting visits and costs of general clinics, specialist clinics, hospitals, Chinese medical doctors, psychologists, and other public and private health units in the past three months. Total expenditure of medical consumption will be calculated.
Quality of life - Short-Form Six Dimensions Health Survey (SF-6D) | at baseline, 3rd, and 6th month
  It is a 6-item survey to assess health-related quality of life valued by the standard gamble technique. The six-dimension composed of six dimensions of health namely physical functioning, role limitation, social functioning, bodily pain, mental health, and vitality. The quality-adjusted life-year (QALY) and the preference-based utility value of the health state can be estimated using a scoring algorithm validated for the Chinese Hong Kong population.
Well-being - PERMA-Profiler (PERMA) | at baseline, 3rd, and 6th month
  It includes 23 items to assess well-being of respondents using a 11-point Likert scale from 0 (never/terrible/not at all) to 10 (always/excellent/completely). Average scores will be calculated, with high scores indicate better well-being. It includes domains in positive emotion, engagement, relationship, meaning, accomplishment, negative emotion, physical health, loneliness, and overall well-being.
Workplace well-being | at baseline, 3rd, and 6th month
  It includes 24 items to examine respondents' well-being in workplace using 6-point Likert scale from 1 (never/strongly disagree) to 7 (always/strongly agree). It includes domains in support from colleagues & company, emotional and work-life balance, gains from job, mental health resources, and company culture. Average scores will be calculated, with high scores indicate better workplace well-being.
Treatment acceptability | at baseline, 3rd, and 6th month
  It includes 4 items to examine the overall user satisfaction toward the online mental health platform. Average scores will be calculated, with high scores indicate higher levels of treatment acceptability.
Implicit Theories of Intelligence (Self-Theory Scale) | at baseline, 3rd, and 6th month
  It includes 8 items to examine respondents' beliefs on whether they can change their mental well-being by making efforts using 6-point Likert scale from 1 (strongly agree) to 6 (strongly disagree). The Cronbach's alpha was 0.9.
Self-Efficacy - General Self-Efficacy Scale (GSE-6) | at baseline, 3rd, and 6th month
  Short form of the General Self-Efficacy Scale (GSE-6). It was developed based on the full General Self-Efficacy Scale (GSE). It includes 6 items with the highest coefficients of variation in GSE to assess respondents' self-efficacy using 4-point scale from 1 (not at all trye) to 4 (exactly true). The Cronbach's alpha was 0.79 to 0.88.
Resilience - Connor-Davidson Resilience Scale (CD-RISC-2) | at baseline, 3rd, and 6th month
  It includes 2 items to measure respondents' stress coping ability using 5-point Likert scale from 0 (never) to 4 (always). Total scores will be calculated. It ranges from 0 to 8, with high scores indicate higher levels in resilience.
Nonattachment - Nonattachment Scale-Short Form (NAS-SF) | at baseline, 3rd, and 6th month
  It includes 8 items to measure nonattachment using 6-point Likert scale from 1 (strongly disagree) to 6 (strongly agree). Average scores will be calculated, with high scores indicate higher levels of nonattachment.
Emotion Regulation - Emotion Regulation Questionnaire (ERQ) | at baseline, 3rd, and 6th month
  It includes 10 items to measure respondents' approach in regulating their emotion using 7-point Likert scale from 0 (strongly disagree) to 7 (strongly agree). Average scores will be calculated, with high scores indicate higher levels of emotion regulation
Work and Social Adjustment - Work and Social Adjustment (WSAS) | at baseline, 3rd, and 6th month
  It includes 5 items to measure participants perceived functional impairment using a 9-point Likert scale from 0 (not at all impaired) to 8 (very severely impaired). Total scores range from 0 to 40, with high scores indicate higher levels of functional impairment.
Daily Hassles - LIVES-Daily Hassles Scale (LIVES-DHS) | at baseline, 3rd, and 6th month
  It measure the extent to which a series of potential daily hassles concern participants using a 5-point Likert scale from 1 (not at all) to 5 (very much). Average scores will be calculated, with high scores indicate higher levels of concerns in potential daily hassles. The scale consists of 18 items to evaluate five sources of daily hassles, included professional, environmental, relational, physical and financial.
Attitude towards Psychological Online Intervention (APOI) | at baseline, 3rd, and 6th month
  It measures respondents' attitude towards psychological online intervention using a 5-point Likert scale from 1 (strongly agree) to 5 (strongly disagree). The scale consists of 16 items to evaluate participants' attitude towards scepticism and perception of risks, confidence in effectiveness, technologization threat, and anonymity benefits in psychological online intervention.
Behavioural Intention - E-therapy Attitude and Process Questionnaire (eTAP) | at baseline, 3rd, and 6th month
  It includes 3 items to measures participants' intention in using online psychological intervention. It is measured by a 7-point Likert scale from 1 (strongly disagree) to 7 (strongly agree) . The subscale showed excellence reliability (Cronbach's alpha = 0.94).
Subjective Norm - E-therapy Attitude and Process Questionnaire (eTAP) | at baseline, 3rd, and 6th month
  It includes 4 items to measures the subjective norm towards online psychological intervention using a 7-point Likert scale from 1 (strongly disagree) to 7 (strongly agree). Three items were adapted in the context of Hong Kong. Two relevant items were constructed and included in the scale. They are 'people in my social network will use online interventions if they have mental health needs' and 'people in my social network world support using online interventions for mental health'.
Mental Health Experiences - The Mental Health Experiences Questionnaire | at baseline, 3rd, and 6th month
  The Mental Health Experiences Questionnaire measures whether respondents access mental health services by 9 items. One question regarding the mode of mental health service or related resources is added. Moreover, options are adapted in the context of Hong Kong. For example, in the question regarding the accessed service and resources, respondents can choose from workshop, group, and one-on-one therapy as they are common resources in Hong Kong.
Self-Stigma - The Self-Stigma of Seeking Psychological Help (SSOSH) | at baseline, 3rd, and 6th month
  It measures the reaction of respondents when they seek help from mental health professionals. This is measured by 10 items using 5-point Likert scale from 1 (strongly disagree) to 7 (strongly agree).
Coping strategy - The Proactive Coping Inventory (PCI) | at baseline, 3rd, and 6th month
  It includes 7 domains and this study only includes 5 domains from the scale, which measure proactive coping, strategic planning, instrumental support seeking, emotional support seeking, and avoidance coping. Coping strategy is measured by thirty-four items using a 4-points scale from 1 (not at all true) to 4 (completely true) in this study
Tolerance for Ambiguity - Tolerance for Ambiguity Scale (TAS) | at baseline, 3rd, and 6th month
  It consists of 12 items to measure respondents' tendency to perceive ambiguous situation as desirable using 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree). Research found improved internal consistency and factor structure for TAS compared to common measure of tolerance for ambiguity in existing literature.
System Usability - System Usability Scale | at baseline, 3rd, and 6th month
  It consists of 10 items to measure the experience of using the online platform. It is a 5-point Likert scale from 0 (strongly disagree) to 4 (strongly agree). To calculate SUS score, item scores of each respondent are summed up and then multiplied by 2.5. The range of score is 0 to 100. A SUS score above 68 would be considered as above average
Work Engagement - Utrecht Work Engagement Scale (UWES-3) | at baseline, 3rd, and 6th month
  It includes 3 items to measure participants experience of being engaged at work in 7-point Likert scale from 0 (Never) to 6 (always/everyday). It shared 86-92% variance with longer nine-item version and pattern of correlation of both versions was similar

CONTACTS AND LOCATIONS:
Locations (1):
- Diversity and Well-being Lab, CUHK, Shatin, N.T., Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Abd-Alrazaq AA, Alajlani M, Alalwan AA, Bewick BM, Gardner P, Househ M. An overview of the features of chatbots in mental health: A scoping review. Int J Med Inform. 2019 Dec;132:103978. doi: 10.1016/j.ijmedinf.2019.103978. Epub 2019 Sep 25. PMID 31622850
- [Background] Andrews G, Basu A, Cuijpers P, Craske MG, McEvoy P, English CL, Newby JM. Computer therapy for the anxiety and depression disorders is effective, acceptable and practical health care: An updated meta-analysis. J Anxiety Disord. 2018 Apr;55:70-78. doi: 10.1016/j.janxdis.2018.01.001. Epub 2018 Feb 1. PMID 29422409
- [Background] Araya R, Flynn T, Rojas G, Fritsch R, Simon G. Cost-effectiveness of a primary care treatment program for depression in low-income women in Santiago, Chile. Am J Psychiatry. 2006 Aug;163(8):1379-87. doi: 10.1176/ajp.2006.163.8.1379. PMID 16877650
- [Background] Ayse, E. B. (2018). Adaptation of the PERMA Well-Being Scale into Turkish: Validity and reliability Studies. Educational Research and Reviews, 13(4), 129-35.
- [Background] Bouwmans, C., Hakkaart-van Roijen, L., Koopmanschap, M., Krol, M., Severens, H., Brouwer, W. (2013). Manual of the iMTA Productivity Cost Questionnaire (iPCQ). Rotterdam: iMTA, Erasmus University Rotterdam.
- [Background] Bouwmans C, Krol M, Brouwer W, Severens JL, Koopmanschap MA, Hakkaart L. IMTA Productivity Cost Questionnaire (IPCQ). Value Health. 2014 Nov;17(7):A550. doi: 10.1016/j.jval.2014.08.1791. Epub 2014 Oct 26. No abstract available. PMID 27201788
- [Background] Bower P, Gilbody S. Stepped care in psychological therapies: access, effectiveness and efficiency. Narrative literature review. Br J Psychiatry. 2005 Jan;186:11-7. doi: 10.1192/bjp.186.1.11. PMID 15630118
- [Background] Brazier J, Usherwood T, Harper R, Thomas K. Deriving a preference-based single index from the UK SF-36 Health Survey. J Clin Epidemiol. 1998 Nov;51(11):1115-28. doi: 10.1016/s0895-4356(98)00103-6. PMID 9817129
- [Background] Briggs AH, Wonderling DE, Mooney CZ. Pulling cost-effectiveness analysis up by its bootstraps: a non-parametric approach to confidence interval estimation. Health Econ. 1997 Jul-Aug;6(4):327-40. doi: 10.1002/(sici)1099-1050(199707)6:43.0.co;2-w. PMID 9285227
- [Background] Butler, J., & Kern, M. L. (2016). The PERMA-Profiler: A brief multidimensional measure of flourishing. International Journal of Wellbeing, 6(3), 1-48.
- [Background] Buttorff C, Hock RS, Weiss HA, Naik S, Araya R, Kirkwood BR, Chisholm D, Patel V. Economic evaluation of a task-shifting intervention for common mental disorders in India. Bull World Health Organ. 2012 Nov 1;90(11):813-21. doi: 10.2471/BLT.12.104133. Epub 2012 Sep 14. PMID 23226893
- [Background] Choi I, Andrews G, Sharpe L, Hunt C. Help-seeking characteristics of Chinese- and English-speaking Australians accessing Internet-delivered cognitive behavioural therapy for depression. Soc Psychiatry Psychiatr Epidemiol. 2015 Jan;50(1):89-97. doi: 10.1007/s00127-014-0956-3. Epub 2014 Sep 6. PMID 25193374
- [Background] Choi I, Zou J, Titov N, Dear BF, Li S, Johnston L, Andrews G, Hunt C. Culturally attuned Internet treatment for depression amongst Chinese Australians: a randomised controlled trial. J Affect Disord. 2012 Feb;136(3):459-68. doi: 10.1016/j.jad.2011.11.003. Epub 2011 Dec 16. PMID 22177742
- [Background] City Mental Health Alliance Hong Kong. (2018). The cost of mental ill health for employers in Hong Kong. Hong Kong: City Mental Health Alliance Hong Kong.
- [Background] City Mental Health Alliance Hong Kong. (2019). Mental health in the workplace: Survey of Hong Kong employees in professional services firms. Hong Kong: City Mental Health Alliance Hong Kong.
- [Background] Czabala C, Charzynska K, Mroziak B. Psychosocial interventions in workplace mental health promotion: an overview. Health Promot Int. 2011 Dec;26 Suppl 1:i70-84. doi: 10.1093/heapro/dar050. PMID 22079937
- [Background] DaPonte, D., Talbot, F., Titov, N., Dear, B. F., Hadjistavropoulos, H. D., Hadjistavropoulos, T., & Jbilou, J. (2018). Facilitating the dissemination of iCBT for the treatment of anxiety and depression: A feasibility study. Behaviour Change, 35(3), 139-151.
- [Background] Dorow M, Lobner M, Pabst A, Stein J, Riedel-Heller SG. Preferences for Depression Treatment Including Internet-Based Interventions: Results From a Large Sample of Primary Care Patients. Front Psychiatry. 2018 May 17;9:181. doi: 10.3389/fpsyt.2018.00181. eCollection 2018. PMID 29867605
- [Background] Dube P, Kurt K, Bair MJ, Theobald D, Williams LS. The p4 screener: evaluation of a brief measure for assessing potential suicide risk in 2 randomized effectiveness trials of primary care and oncology patients. Prim Care Companion J Clin Psychiatry. 2010;12(6):PCC.10m00978. doi: 10.4088/PCC.10m00978blu. PMID 21494337
- [Background] Fitzpatrick KK, Darcy A, Vierhile M. Delivering Cognitive Behavior Therapy to Young Adults With Symptoms of Depression and Anxiety Using a Fully Automated Conversational Agent (Woebot): A Randomized Controlled Trial. JMIR Ment Health. 2017 Jun 6;4(2):e19. doi: 10.2196/mental.7785. PMID 28588005
- [Background] Gerhards SA, de Graaf LE, Jacobs LE, Severens JL, Huibers MJ, Arntz A, Riper H, Widdershoven G, Metsemakers JF, Evers SM. Economic evaluation of online computerised cognitive-behavioural therapy without support for depression in primary care: randomised trial. Br J Psychiatry. 2010 Apr;196(4):310-8. doi: 10.1192/bjp.bp.109.065748. PMID 20357309
- [Background] Giangrasso, B. (2018). Psychometric properties of the PERMA-Profiler as hedonic and eudaimonic well-being measure in an Italian context. Current Psychology, 40, 1-10.
- [Background] Gross JJ, John OP. Individual differences in two emotion regulation processes: implications for affect, relationships, and well-being. J Pers Soc Psychol. 2003 Aug;85(2):348-62. doi: 10.1037/0022-3514.85.2.348. PMID 12916575
- [Background] Hedman E, Ljotsson B, Lindefors N. Cognitive behavior therapy via the Internet: a systematic review of applications, clinical efficacy and cost-effectiveness. Expert Rev Pharmacoecon Outcomes Res. 2012 Dec;12(6):745-64. doi: 10.1586/erp.12.67. PMID 23252357
- [Background] Ho FY, Yeung WF, Ng TH, Chan CS. The Efficacy and Cost-Effectiveness of Stepped Care Prevention and Treatment for Depressive and/or Anxiety Disorders: A Systematic Review and Meta-Analysis. Sci Rep. 2016 Jul 5;6:29281. doi: 10.1038/srep29281. PMID 27377429
- [Background] Hollinghurst S, Peters TJ, Kaur S, Wiles N, Lewis G, Kessler D. Cost-effectiveness of therapist-delivered online cognitive-behavioural therapy for depression: randomised controlled trial. Br J Psychiatry. 2010 Oct;197(4):297-304. doi: 10.1192/bjp.bp.109.073080. PMID 20884953
- [Background] Iasiello, M., Bartholomaeus, J., Jarden, A., & Kelly, G. (2017). Measuring PERMA+ in South Australia, the State of Wellbeing: A comparison with national and international norms. Journal of Positive Psychology and Wellbeing, 1(2), 53-72.
- [Background] Khaw, D., & Kern, M. (2014). A cross-cultural comparison of the PERMA model of well-being. Undergraduate Journal of Psychology at Berkeley, University of California, 8, 10-23.
- [Background] Katon WJ, Schoenbaum M, Fan MY, Callahan CM, Williams J Jr, Hunkeler E, Harpole L, Zhou XH, Langston C, Unutzer J. Cost-effectiveness of improving primary care treatment of late-life depression. Arch Gen Psychiatry. 2005 Dec;62(12):1313-20. doi: 10.1001/archpsyc.62.12.1313. PMID 16330719
- [Background] Kleiboer A, Donker T, Seekles W, van Straten A, Riper H, Cuijpers P. A randomized controlled trial on the role of support in Internet-based problem solving therapy for depression and anxiety. Behav Res Ther. 2015 Sep;72:63-71. doi: 10.1016/j.brat.2015.06.013. Epub 2015 Jul 6. PMID 26188373
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Ladapo JA, Shaffer JA, Fang Y, Ye S, Davidson KW. Cost-effectiveness of enhanced depression care after acute coronary syndrome: results from the Coronary Psychosocial Evaluation Studies randomized controlled trial. Arch Intern Med. 2012 Nov 26;172(21):1682-4. doi: 10.1001/archinternmed.2012.4448. No abstract available. PMID 23070196
- [Background] Lam CL, Brazier J, McGhee SM. Valuation of the SF-6D Health States Is Feasible, Acceptable, Reliable, and Valid in a Chinese Population. Value Health. 2008 Mar-Apr;11(2):295-303. doi: 10.1111/j.1524-4733.2007.00233.x. PMID 18380642
- [Background] Lam LC, Wong CS, Wang MJ, Chan WC, Chen EY, Ng RM, Hung SF, Cheung EF, Sham PC, Chiu HF, Lam M, Chang WC, Lee EH, Chiang TP, Lau JT, van Os J, Lewis G, Bebbington P. Prevalence, psychosocial correlates and service utilization of depressive and anxiety disorders in Hong Kong: the Hong Kong Mental Morbidity Survey (HKMMS). Soc Psychiatry Psychiatr Epidemiol. 2015 Sep;50(9):1379-88. doi: 10.1007/s00127-015-1014-5. Epub 2015 Feb 8. PMID 25660760
- [Background] Mak WW, Chan AT, Cheung EY, Lin CL, Ngai KC. Enhancing Web-based mindfulness training for mental health promotion with the health action process approach: randomized controlled trial. J Med Internet Res. 2015 Jan 19;17(1):e8. doi: 10.2196/jmir.3746. PMID 25599904
- [Background] Mak WW, Chio FH, Chan AT, Lui WW, Wu EK. The Efficacy of Internet-Based Mindfulness Training and Cognitive-Behavioral Training With Telephone Support in the Enhancement of Mental Health Among College Students and Young Working Adults: Randomized Controlled Trial. J Med Internet Res. 2017 Mar 22;19(3):e84. doi: 10.2196/jmir.6737. PMID 28330831
- [Background] Mak WW, Tong AC, Yip SY, Lui WW, Chio FH, Chan AT, Wong CC. Efficacy and Moderation of Mobile App-Based Programs for Mindfulness-Based Training, Self-Compassion Training, and Cognitive Behavioral Psychoeducation on Mental Health: Randomized Controlled Noninferiority Trial. JMIR Ment Health. 2018 Oct 11;5(4):e60. doi: 10.2196/mental.8597. PMID 30309837
- [Background] Mulhern B, Mukuria C, Barkham M, Knapp M, Byford S, Soeteman D, Brazier J. Using generic preference-based measures in mental health: psychometric validity of the EQ-5D and SF-6D. Br J Psychiatry. 2014 Sep;205(3):236-43. doi: 10.1192/bjp.bp.112.122283. Epub 2014 May 22. PMID 24855127
- [Background] National Institute for Health and Clinical Excellence (NICE) (2006). Computerized cognitive behaviour therapy for depression and anxiety. London: National Institute for Health and Clinical Excellence.
- [Background] Ni MY, Li TK, Yu NX, Pang H, Chan BH, Leung GM, Stewart SM. Normative data and psychometric properties of the Connor-Davidson Resilience Scale (CD-RISC) and the abbreviated version (CD-RISC2) among the general population in Hong Kong. Qual Life Res. 2016 Jan;25(1):111-6. doi: 10.1007/s11136-015-1072-x. Epub 2015 Jul 22. PMID 26198665
- [Background] NICE Guidance. (2018). Common mental health problems: Identification and pathways to care. Retrieved from https://www.nice.org.uk/guidance/cg123/resources/common-mental-health-problems-identification-and-pathways-to-care-pdf-35109448223173
- [Background] Romero C, Master A, Paunesku D, Dweck CS, Gross JJ. Academic and emotional functioning in middle school: the role of implicit theories. Emotion. 2014 Apr;14(2):227-34. doi: 10.1037/a0035490. Epub 2014 Feb 10. PMID 24512251
- [Background] Ryan J, Curtis R, Olds T, Edney S, Vandelanotte C, Plotnikoff R, Maher C. Psychometric properties of the PERMA Profiler for measuring wellbeing in Australian adults. PLoS One. 2019 Dec 23;14(12):e0225932. doi: 10.1371/journal.pone.0225932. eCollection 2019. PMID 31869336
- [Background] Schaufeli, W. B., Shimazu, A., Hakanen, J., SALANOVA, M., & WITTE, H. (2017). An Ultra-Short Measure for Work Engagement The UWES-3 Validation Across Five Countries, 1-15, 2017.
- [Background] Schaufeli, W. B., Shimazu, A., Hakanen, J., Salanova, M., & De Witte, H. (2019). An ultra-short measure for work engagement: the UWES-3 validation across five countries. European Journal of Psychological Assessment, 35(4), 577.
- [Background] Schwarzer, R., & Jerusalem, M. (1995). Generalized Self-Efficacy scale. In J. Weinman, S. Wright, & M. Johnston, Measures in health psychology: A user's portfolio. Causal and control beliefs (pp. 35-37). Windsor, UK: NFER-NELSON.
- [Background] Schwarzer, R., Bäßler, J., Kwiatek, P., Schröder, K., & Zhang, J. X. (1997). The assessment of optimistic self-beliefs: Comparison of the German, Spanish, and Chinese versions of the general self-efficacy scale. Applied Psychology, 46(1), 69-88.
- [Background] Simon GE, Katon WJ, Lin EH, Rutter C, Manning WG, Von Korff M, Ciechanowski P, Ludman EJ, Young BA. Cost-effectiveness of systematic depression treatment among people with diabetes mellitus. Arch Gen Psychiatry. 2007 Jan;64(1):65-72. doi: 10.1001/archpsyc.64.1.65. PMID 17199056
- [Background] Sit, R. W. S. (2019). Clinical effectiveness of hypertonic dextrose prolotherapy in chronic ankle instability: A randomized clinical trial. School of Public Health, CUHK. Unpublished.
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Titov N, Andrews G, Johnston L, Robinson E, Spence J. Transdiagnostic Internet treatment for anxiety disorders: A randomized controlled trial. Behav Res Ther. 2010 Sep;48(9):890-9. doi: 10.1016/j.brat.2010.05.014. Epub 2010 May 24. PMID 20561606
- [Background] Titov N, Dear BF, Johnston L, Lorian C, Zou J, Wootton B, Spence J, McEvoy PM, Rapee RM. Improving adherence and clinical outcomes in self-guided internet treatment for anxiety and depression: randomised controlled trial. PLoS One. 2013 Jul 3;8(7):e62873. doi: 10.1371/journal.pone.0062873. Print 2013. PMID 23843932
- [Background] Udayar S, Urbanaviciute I, Morselli D, Bollmann G, Rossier J, Spini D. The LIVES Daily Hassles Scale and Its Relation to Life Satisfaction. Assessment. 2023 Mar;30(2):348-363. doi: 10.1177/10731911211047894. Epub 2021 Oct 18. PMID 34663113
- [Background] Vaishnavi S, Connor K, Davidson JR. An abbreviated version of the Connor-Davidson Resilience Scale (CD-RISC), the CD-RISC2: psychometric properties and applications in psychopharmacological trials. Psychiatry Res. 2007 Aug 30;152(2-3):293-7. doi: 10.1016/j.psychres.2007.01.006. Epub 2007 Apr 25. PMID 17459488
- [Background] van Straten A, Hill J, Richards DA, Cuijpers P. Stepped care treatment delivery for depression: a systematic review and meta-analysis. Psychol Med. 2015 Jan;45(2):231-46. doi: 10.1017/S0033291714000701. Epub 2014 Mar 26. PMID 25065653
- [Background] Wang, L., Ding, R., Hu, D., & Li, S. (2014). The value of Chinese version GAD-7 and PHQ-9 to screen anxiety and depression in cardiovascular outpatients. Journal of American College of Cardiology, 64(16_S), C222.
- [Background] Zahra D, Qureshi A, Henley W, Taylor R, Quinn C, Pooler J, Hardy G, Newbold A, Byng R. The work and social adjustment scale: reliability, sensitivity and value. Int J Psychiatry Clin Pract. 2014 Jun;18(2):131-8. doi: 10.3109/13651501.2014.894072. Epub 2014 Mar 16. PMID 24527886
- [Background] Brooke, J. (1996). SUS-A quick and dirty usability scale. Usability evaluation in industry, 189(194), 4-7.
- [Background] Clough BA, Eigeland JA, Madden IR, Rowland D, Casey LM. Development of the eTAP: A brief measure of attitudes and process in e-interventions for mental health. Internet Interv. 2019 Jun 18;18:100256. doi: 10.1016/j.invent.2019.100256. eCollection 2019 Dec. PMID 31890610
- [Background] De Castella, K., & Byrne, D. (2015). My intelligence may be more malleable than yours: The revised implicit theories of intelligence (self-theory) scale is a better predictor of achievement, motivation, and student disengagement. European Journal of Psychology of Education, 30(3), 245-267.
- [Background] Greenglass, E., Schwarzer, R., Jakubiec, D., Fiksenbaum, L., & Taubert, S. (1999). The proactive coping inventory (PCI): A multidimensional research instrument. In 20th international conference of the stress and anxiety research society (STAR), Cracow, Poland (Vol. 12, p. 14).
- [Background] Herman, J. L., Stevens, M. J., Bird, A., Mendenhall, M., & Oddou, G. (2010). The tolerance for ambiguity scale: Towards a more refined measure for international management research. International Journal of Intercultural Relations, 34(1), 58-65.
- [Background] Patten SB, Williams JV, Lavorato DH, Bulloch AG, Charbonneau M, Gautam M, Moss P, Abbey S, Stuart H. Perceived Stigma among Recipients of Mental Health Care in the General Canadian Population. Can J Psychiatry. 2016 Aug;61(8):480-8. doi: 10.1177/0706743716639928. Epub 2016 Mar 18. PMID 27310227
- [Background] Romppel M, Herrmann-Lingen C, Wachter R, Edelmann F, Dungen HD, Pieske B, Grande G. A short form of the General Self-Efficacy Scale (GSE-6): Development, psychometric properties and validity in an intercultural non-clinical sample and a sample of patients at risk for heart failure. Psychosoc Med. 2013;10:Doc01. doi: 10.3205/psm000091. Epub 2013 Feb 20. PMID 23429426
- [Background] Schroder J, Sautier L, Kriston L, Berger T, Meyer B, Spath C, Kother U, Nestoriuc Y, Klein JP, Moritz S. Development of a questionnaire measuring Attitudes towards Psychological Online Interventions-the APOI. J Affect Disord. 2015 Nov 15;187:136-41. doi: 10.1016/j.jad.2015.08.044. Epub 2015 Aug 28. PMID 26331687
- [Background] Vogel, D. L., Wade, N. G., & Haake, S. (2006). Measuring the self-stigma associated with seeking psychological help. Journal of counseling psychology, 53(3), 325.